CLINICAL TRIAL: NCT06770088
Title: A Prospective, Single-arm, Multicenter Study to Explore the Efficacy and Safety of Vunakizumab in Adults with Active Spondyloarthritis
Brief Title: Vunakizumab in Adults with Spondyloarthritis
Acronym: V SPA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-371-01
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Spondyloarthritis (SpA)
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Active Comparator): Vunakizumab
  Interventions: Drug: vnacicizumab

INTERVENTIONS:
Drug: vnacicizumab — Vunakizumab 120 mg subcutaneous injection at baseline and week2, week4, then every other 4 weeks.

SUMMARY:
This prospective, single-arm, multicenter study is aimed to explore the efficacy and safety of Vunakizumab in adults with spondyloarthritis. The primary endpoint is the proportion of adults with spondyloarthritis achieving ankylosing spondylitis assessment score (ASAS) 40 at week 16 in the treatment of Vunakizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years when signing the informed consent;
2. Patients diagnosed with spondyloarthritis (excluding psoriatic arthritis) and are eligible for biologic therapy;
3. The subjects voluntarily signed informed consent before the start of any procedures related to the study, were able to communicate with the investigators smoothly, understood and were willing to strictly abide by the requirements of the clinical research protocol to complete the study.

Exclusion Criteria:

1. Patients with severe hypersensitivity reaction to the active ingredient or any excipient of Vunakizumab;
2. fertile women (defined as all women with the physical requirements for pregnancy) and men who are pregnant or who are unwilling or unable to use highly effective birth control during the study and within 20 weeks after last receiving the study drug;
3. active infection with important clinical significance;
4. patients with moderate to severe heart failure (NYHA class Ⅲ/Ⅳ);
5. patients with malignant tumors who were receiving treatment or were not receiving treatment;
6. concomitant with other inflammatory diseases or severe autoimmune diseases, including but not limited to inflammatory bowel disease, which may affect the efficacy and safety evaluation according to the investigator's judgment;
7. any other condition that the investigator considers would prevent the subject from adhering to and completing the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with spondyloarthritis who achieved ASAS40 response | week 16
  Proportion of patients with spondyloarthritis who achieved ASAS40 response

SECONDARY OUTCOMES:
The proportion of patients achieving ASAS20 | Week 16
  The proportion of patients achieving ASAS20
Proportion of patients with spondyloarthritis who achieved ASAS20 response | Week 52
  Proportion of patients with spondyloarthritis who achieved ASAS20 response

IPD SHARING:
Plan to Share IPD: Undecided